CLINICAL TRIAL: NCT02134834
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, Single Dose Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of OP0595 Administered Intravenously in Healthy Male Subjects.
Brief Title: A Phase I Study to Assess Safety, Tolerability and Pharmacokinetics of OP0595
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Meiji Seika Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OP0595-1
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2014-12-12 (Estimated); Status verified 2014-12

CONDITIONS: Healthy Volunteers; Bacterial Infections
MeSH Terms: conditions — Bacterial Infections | interventions — nacubactam

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ascending single dose of OP0595 (Experimental)
  Interventions: Drug: OP0595
- Normal Saline (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: OP0595 — Five cohorts of 8 subjects (6 active and 2 placebo) are planned for evaluation
  Arms: Ascending single dose of OP0595
Drug: Placebo — Five cohorts of 8 subjects (6 active and 2 placebo) are planned for evaluation
  Arms: Normal Saline

SUMMARY:
The objectives of this study are to assess the safety, tolerability and pharmacokinetic profile of OP0595 administered intravenously to healthy male, Caucasian, adult subjects at single escalating doses.

ELIGIBILITY:
Inclusion Criteria:

* Caucasian males aged between 18 and 45 years (inclusive) at Screening
* A Body Mass Index (BMI) between 18.0 and 30.0 kg/m² (inclusive) at Screening
* Good general health as determined by the Investigator based on medical history, physical examination, vital signs, 12-lead ECG and clinical laboratory tests
* Negative urine test for drugs of abuse and breath test for alcohol both at Screening and Day -1

Exclusion Criteria:

* Receipt of any investigational agent or drug within four months before Screening
* A history or current evidence of allergic symptoms such as bronchial asthma, drug-induced rash or urticaria
* Hypersensitivity and/or allergy to drugs
* Concurrent or history of clinically significant cardiovascular, hepatic, renal, endocrine, gastrointestinal, respiratory, psychiatric, neurologic and/or hematological disorders
* A history of chronic or recurrent infections or current active infection
* A recent history of surgery within three months prior to Screening, determined by the Investigator to be clinically relevant
* A history or presence of malignancy
* Donation of blood (or loss of blood) greater than 400 ml within three months before Screening
* A history of smoking at any time within one year before Screening

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-05; Primary Completion 2014-08 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Safety from baseline through the end of the study | Day 1 to Day 7
  Number of patients with adverse events

SECONDARY OUTCOMES:
Plasma PK parameters of OP0595 and its metabolites | Day 1 to Day 2
  Cmax, tmax, AUC0-last, AUC0-inf, Kel, T1/2, CLtot, Vdss
Urine PK parameters of OP0595 and its metabolites | Day 1 to Day 2
  Ae, Ae0-t, Ae0-t/Dose, CLr

CONTACTS AND LOCATIONS:
Overall Officials: Mitsuharu Egawa, Study Chair — Meiji Seika Pharma Co., Ltd.
Locations (1):
- Perth, Western Australia, Australia

REFERENCES:
- [Derived] Mallalieu NL, Winter E, Fettner S, Patel K, Zwanziger E, Attley G, Rodriguez I, Kano A, Salama SM, Bentley D, Geretti AM. Safety and Pharmacokinetic Characterization of Nacubactam, a Novel beta-Lactamase Inhibitor, Alone and in Combination with Meropenem, in Healthy Volunteers. Antimicrob Agents Chemother. 2020 Apr 21;64(5):e02229-19. doi: 10.1128/AAC.02229-19. Print 2020 Apr 21. PMID 32041717